CLINICAL TRIAL: NCT00758914
Title: Vitamin E and Infection in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Simin Nikbin Meydani, DVM, PhD, Tufts University
Other Study IDs: 1R01AG013975 (NIH)
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Respiratory Infection; Elderly
Keywords: Vitamin E
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Vitamin E — 200 IU alpha-tocopherol or placebo for 1 year.

SUMMARY:
Aging is associated with a variety of changes in the immune system. These changes result in a less effective immune response, which places the elderly at a greater risk for infection and disease. Respiratory infections cause a great number of morbidity and mortality in the elderly population. Vitamin E has been known to improve the immune response of the elderly and has been suggested for use in preventative strategies for this population. The purpose of this study is to examine the effect of one year vitamin supplementation on respiratory infection in the elderly population residing in nursing homes. This study was conducted using a randomized, double blind, placebo controlled clinical trial at 33 long-term care facilities in the greater Boston area. A total of 617 subjects over the age of 65 were enrolled in the study, with 451 completers. The participants were supplemented wit either 200 IU of vitamin E per day or placebo. The primary outcomes consisted of respiratory tract infection, number of sick days, and antibiotic use. The study involved use of questionnaires, standard anthropometrics measurements, non-invasive body composition, blood and urine sample collection, and delayed type test (DTH) using the Mantoux method. This study has been closed since August 2000 and is in the stage of data analysis only.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older;
* life expectancy greater than 6 months;
* no anticipated discharge within 3 months;
* not room-bound for the past 3 months;
* absence of active neoplastic disease;
* no tube feeding, no kidney dialysis;
* no intravenous or urethral catheters for the last 30 days;
* no tracheostomy or chronic ventilator;
* antibiotic-free for more than 2 weeks;
* no long-term steroid treatment greater than 10 mg/d, no use of immunosuppressive drugs, or greater than the recommended daily allowance (RDA) level of supplements of vitamins E, C, or B6, selenium, zinc, beta-carotene, or fish oil;
* body mass index of at least 18;
* serum albumin at least 3.0 g/dL; able to swallow pills;
* willing to receive influenza vaccine;
* willing to provide informed consent (for patients with dementia, family members provided informed consent)

Exclusion Criteria:

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Start 1997-05; Primary Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Belisle SE, Hamer DH, Leka LS, Dallal GE, Delgado-Lista J, Fine BC, Jacques PF, Ordovas JM, Meydani SN. IL-2 and IL-10 gene polymorphisms are associated with respiratory tract infection and may modulate the effect of vitamin E on lower respiratory tract infections in elderly nursing home residents. Am J Clin Nutr. 2010 Jul;92(1):106-14. doi: 10.3945/ajcn.2010.29207. Epub 2010 May 19. PMID 20484443